CLINICAL TRIAL: NCT00919997
Title: HPV Infection in Indian HIV-Seropositive Men Who Have Sex With Men (MSM)
Brief Title: Human Papilloma Virus Infection in HIV-Positive Indian Men Who Have Sex With Men
Status: Completed | Type: Observational
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: AMC-060; U01CA121947 (NIH); CDR0000629624 (Other: NCI)
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Nonneoplastic Condition; Precancerous Condition
Keywords: human papilloma virus infection; HIV infection; HIV Infections
MeSH Terms: conditions — Precancerous Conditions; Papillomavirus Infections; HIV Infections | interventions — Polymerase Chain Reaction; Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Anal cytology Penile cytology Saliva Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Specimen collection: Single group study. Blood, saliva, anal cytology, and penile cytology samples, and questionnaire responses will be collected from participants at a single study visit.
  Interventions: Genetic: DNA analysis; Genetic: polymerase chain reaction; Other: fluorescence activated cell sorting; Other: questionnaire administration; Other: study of socioeconomic and demographic variables; Procedure: study of high risk factors

INTERVENTIONS:
Genetic: DNA analysis — Anal pap smear, penile pap smear, blood collection, and saliva collection at a single study visit for HPV DNA analysis.
Genetic: polymerase chain reaction — Blood and saliva samples collected at a single study visit will be analyzed for for HPV DNA.
Other: fluorescence activated cell sorting — Blood and saliva samples collected at a single study visit will be analyzed for for HPV DNA.
Other: questionnaire administration — Describe risk factors for penile, anal and oral HPV infection in Indian HIV-seropositive MSM.
Other: study of socioeconomic and demographic variables — Describe risk factors for penile, anal and oral HPV infection in Indian HIV-seropositive MSM.
Procedure: study of high risk factors — Describe risk factors for penile, anal and oral HPV infection in Indian HIV-seropositive MSM.

SUMMARY:
RATIONALE: Gathering information about human papilloma virus (HPV) infection in HIV-positive men who have sex with men may help doctors learn more about the disease.

PURPOSE: This clinical trial is studying HPV infection in HIV-positive Indian men who have sex with men.

DETAILED DESCRIPTION:
OBJECTIVES:

* Describe the prevalence of penile, anal, and oral human papilloma virus (HPV) infection in HIV-seropositive Indian men who have sex with men.
* Determine the spectrum of HPV types at these anatomic sites in these patients.
* Determine the distribution of strain variants of HPV 16, 18, and 31 at these anatomic sites in these patients.
* Describe risk factors for penile, anal, and oral HPV infection in these patients.

OUTLINE: This is a multicenter study.

Patients complete interviewer-administered questionnaires on demographics, native place, socioeconomic status, medical history, numbers of sexual partners and sexual practices, circumcision status, and risk factors for oral malignancies and human papilloma virus (HPV), including oral sex, smoking or chewing tobacco, drug use, oral hygiene, and tooth loss.

Patients undergo cell sample collection from the penis, scrotum, anus, and mouth, and saliva sample collection for HPV DNA testing by PCR. Patients also undergo blood sample collection to measure CD4+ count and HIV viral load by FACS and PCR.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* HIV-1 infection, as documented by ELISA and confirmed by a second testing method (e.g., western blot, HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA)

  - If prior documentation and confirmation of HIV-1 infection is not available, two licensed rapid HIV tests are allowed
* Must have had receptive or insertive anal intercourse with another man within the past 6 months

PATIENT CHARACTERISTICS:

* Speaks Hindi (in Mumbai) or Tamil (in Vellore)
* No active drug or alcohol use or dependence that, in the opinion of the site Investigator, would interfere with adherence to study requirements
* No history of a sex-change operation that would preclude collection of penile or scrotal specimens

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1 infected men who have sex with men from Mumbai and Vellore, India, who are age 18 or older.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Detectable human papilloma virus DNA in the penis, anus, or mouth | Study entry

SECONDARY OUTCOMES:
Distribution of strain variants of HPV 16, 18 and 31 | Study entry
Describe risk factors for penile, anal and oral HPV infection in Indian HIV-seropositive MSM | Study entry

CONTACTS AND LOCATIONS:
Overall Officials: Joel Palefsky, MD, Study Chair — University of California, San Francisco; Dilip Mathai, MD, Principal Investigator — Christian Medical College and Hospital; Ashok Row Kavi, Principal Investigator — Humsafar Trust
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States